CLINICAL TRIAL: NCT06081972
Title: Towards a Food Ingredient Clinically Proven to Benefit Gut Health: Novel RG-I Variants
Acronym: NUTRIGUT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Örebro University, Sweden (Other)
Collaborators: NutriLeads B.V. (Wageningen, The Netherlands) (Unknown); ProDigest (Ghent, Belgium) (Unknown); Ambiotis (Toulouse, France) (Unknown)
Responsible Party: Principal Investigator, Robert Brummer, Professor, Örebro University, Sweden
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2023-03938-01
Record Dates: First submitted 2023-09-20; First posted 2023-10-13 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Healthy
Keywords: prebiotic; short - chain fatty acids (SCFAs); Plasmacytoid dendritic cell markers (PDCs); gut microbiota; rhamnogalacturonan I; immune response
MeSH Terms: interventions — maltodextrin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): Participants who will be randomized in the placebo group will receive maltodextrin (500mg/day).
  Interventions: Dietary Supplement: Maltodextrin
- Chicory RG-I (Experimental): Participants who will be randomized in the placebo group will receive Chicory RG-I (500mg/day).
  Interventions: Dietary Supplement: Chicory RG-I
- Carrot RG-I (Experimental): Participants who will be randomized in the placebo group will receive Carrot RG-I (500mg/day).
  Interventions: Dietary Supplement: Carrot RG-I

INTERVENTIONS:
Dietary Supplement: Maltodextrin — During the feeding period (4 weeks) two capsules/ day will be administered to subjects randomized in this group containing placebo powder with a breakfast item on a daily basis.
  Arms: Placebo
Dietary Supplement: Chicory RG-I — During the feeding period (4 weeks) two capsules/ day will be administered to subjects randomized in this group containing chicory RG-I with a breakfast item on a daily basis.
  Arms: Chicory RG-I
Dietary Supplement: Carrot RG-I — During the feeding period (4 weeks) two capsules/ day will be administered to subjects randomized in this group containing carrot RG-I with a breakfast item on a daily basis.
  Arms: Carrot RG-I

SUMMARY:
The aim of this study is to determine, quantify and understand the potential prebiotic effects of RG-I variants via microbiota modulation. The anti-inflammatory potential effects of these variants will also be investigated.

DETAILED DESCRIPTION:
The plant cell wall derived RG-I (from chicory or carrot) and maltodextrin (placebo) in capsuled form will be provided by the food company NutriLeads B.V (Wageningen, The Netherlands), which has run tests of safety of the products and warranties their food grade quality and safety. The administration of RG-I will be done via a human intervention study of parallel arms, randomized, placebo - controlled, double blinded design (proof of concept study).

The dietary fibre from different RG-I sources will be tested for its prebiotic and immunomodulatory potential. Thus, the effects of these fibres on short chain fatty acid (SCFA) profile, microbiota composition, microbiota-associated metabolites and intestinal inflammatory markers will be investigated from fecal material obtained from the study participants.

The dietary fibre from different RG-I sources will be tested for their immunomodulatory and lifestyle related effects. The effects of fibres on immune activation markers will be investigated from blood samples collected from the study participants.

ELIGIBILITY:
Inclusion Criteria:

1. Signed consent prior to any study related procedures
2. Age 18-70 years
3. Willing to abstain from regular consumption of prebiotics/probiotics/synbiotics products or medication known to alter gastrointestinal functions at least 4 weeks prior to the study visits
4. Body mass index (BMI) ≥ 18.5 and ≤ 30.0 kg m-2

Exclusion Criteria:

1. Previous complicated gastrointestinal surgery
2. Presence of gastrointestinal disorder or any disorder which the principal investigator considers to affect the results of the study
3. Current diagnosis of psychiatric disease
4. Current and past diagnosis inflammatory gastrointestinal disease (e.g. Inflammatory Bowel Disease)
5. Systemic use of antibiotics or steroids medications in the last 3 months prior to study visits
6. Frequent use of NSAID (Non-Steroidal Anti Inflammatory Drugs) the last 2 months prior to study visits
7. Abuse of alcohol or drugs
8. Frequent use of laxatives, anti-diarrheal, anti-cholinergic within last 3 months prior to study visits
9. Pregnancy and breast-feeding
10. Vegan dietary habits or consumption of dietary fibers ≥ 25 g per day according to the food frequency questionnaire
11. Smoking or usage of snus within last 3 months prior to study visits
12. No recent weight loss or gain 5% of their normal weight in the last month

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2023-10-02 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Change from baseline to the effect on selected intestinal microbial populations. | The levels of the selected microbial populations will be measured weekly from baseline till the end of the interventional period.(4 weeks period)
  Selected microbial populations will be quantified with quantitative Polymerase Chain Reaction (PCR).
Change from baseline to the effect on the intestinal microbial populations. | The levels of the microbial populations will be measured weekly from baseline till the end of the interventional period.(4 weeks period)
  Microbial populations will be quantified with 16SRNA sequencing.

SECONDARY OUTCOMES:
Change from baseline to the effect on the intestinal microbial populations's metabolic products [i.e. Short-Chain Fatty Acids (SCFA)]. | SCFAs levels will be evaluated at baseline and at the end of the intervention. (4 weeks period)
  SCFAs will be quantified with Gas chromatography.
Change from baseline to the effect on immune system reinforcement. | Immune system reinforcement will be evaluated at baseline and at the end of the intervention. (4 weeks period)
  Plasmacytoid dendritic cells activation will be evaluated with flow cytometry.
Change from baseline to the effect on inflammation. | Inflammation will be evaluated at baseline and at the end of the intervention. (4 weeks period)
  Inflammatory related markers will be quantified by ELISA techniques.
Change from baseline to the effect on exhaled volatile organic compounds levels. | Exhaled volatile organic compounds levels will be evaluated at baseline and at the end of the intervention. (4 weeks period)
  Exhaled volatile organic compounds levels will be evaluated with Thermal Desorption Gas chromatography.
Change from baseline to the effect on fecal metabolomic fingerprinting. | Metabolomic fingerprinting will be evaluated at baseline and at the end of the intervention. (4 weeks period)
  Metabolomic fingerprinting will be evaluated by applying laser assisted Rapid Evaporative Ionisation Mass Spectrometry (LA-REIMS) method on biological material.
Gastrointestinal tolerance of the supplement. | Gastrointestinal symptoms will be evaluated at baseline and at the end of the intervention. (4 weeks period)
  Gastrointestinal health will be evaluated with the use of a 1-day questionnaire consisting of 13 items concerning satiety, abdominal pain, diarrhea, constipation and bloating.The intensity of each parameter will be assessed on a scale of 0-7, where '0' represents absence of symptoms and '7' severe symptoms.
Dietary habits prior to the initiation of the study. | Dietary habits will be measured at baseline prior to the initiation of the study as background information.
  Dietary habits will be evaluated with the use of food frequency questionnaire (FFQ).
Changes from baseline to the effect on physical activity levels. | Physical activity will be evaluated at baseline and at the end of the intervention. (4 weeks period)
  Physical activity will be evaluated with the use of a validated questionnaire. IPAQ consists of 7 items questions concerning the duration and the intensity of physical activity so absolute numerical data will be obtained from it.
Changes from baseline to the effect on quality of life. | Quality of life will be evaluated at baseline and at the end of the intervention. (4 weeks period)
  Quality of life will be evaluated with the use of a validated questionnaire. EQ-5D-5L consists of 5 items concerning mobility, self-care, usual activities, pain/discomfort, anxiety/depression.The overall score from this questionnaire will be calculated by assigning a numerical value to each response level (i.e., 1 for "no problems", 5 for "extreme problems"/"unable to") and summing these values across the five items, resulting in a score from 5 (11,111, no problems on any dimension) to 25 (55,555, extreme problems on all dimensions).

CONTACTS AND LOCATIONS:
Locations (1):
- Campus USÖ, Örebro, Sweden

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-09-20): https://cdn.clinicaltrials.gov/large-docs/72/NCT06081972/Prot_SAP_000.pdf